CLINICAL TRIAL: NCT04296695
Title: The Efficacy and Safety of Biktarvy in Treatment-Naïve Late Presenters With HIV-1 Infection
Brief Title: Biktarvy in Treatment-Naïve Late Presenters With HIV-1 Infection
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Collaborators: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Gilead ISR-CN-18-10596
Record Dates: First submitted 2020-03-03; First posted 2020-03-05 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: HIV-1-infection
Keywords: Biktarvy; HIV-1 infection
MeSH Terms: interventions — bictegravir, emtricitabine, tenofovir alafenamide, drug combination; Tenofovir; efavirenz

STUDY DESIGN:
Intervention Model Description: Non-inferioty or advantage of B/F/TAF comparing with the first line TDF/3TC/EFV for later presenters in China
Masking Description: randomized, multicentered, open-lable RCT, one arm with B/F/TAF and one arm with TDF/3TC/EFV
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- B/F/TAF (Experimental): 50mg/600mg/300mg
  Interventions: Drug: B/F/TAF
- TDF/3TC/EFV (Active Comparator): 300mg/300mg/400mg
  Interventions: Drug: TDF/3TC/EFV

INTERVENTIONS:
Drug: B/F/TAF — randomized, multicentered, open-lable RCT, one arm with B/F/TAF and one arm with TDF/3TC/EFV
  Other Names: Biktarvy
  Arms: B/F/TAF
Drug: TDF/3TC/EFV — TDF/3TC/EFV
  Other Names: Tenofovir /Ravmidine /Efavirenz
  Arms: TDF/3TC/EFV

SUMMARY:
The efficacy and safety of Biktarvy in Treatment-Naïve Late Presenters with HIV-1 Infection

DETAILED DESCRIPTION:
HIV epidemic is still severe in China, the estimated number if PLWH in HIV is around 1.25 million all of China with an increasing trend of new cases. Late presenters with low CD4 T cells and/or with hight viral load should be paid more attention for better treatment and care. As a new combined antiretroviral regimen of integrase inhibitor, B/F/TAF was recently approved in US and European and also in China which needs more real world data in China. Non-inferiority or advantage of B/F/TAF comparing with the first line TDF/3TC/EFV for later presenters in China needs to be explored.

ELIGIBILITY:
Inclusion Criteria:

1.Ability to understand and sign a written informed consent form 2.18 years old or older 3.Confirmed HIV-antibody positive through Western Blot testing without any previous ART 4.CD4 < 200/mm3, VL >1000 copies/ml 5.Estimated glomerular filtration rate (GFR) ≥ 50 mL/min (calculated by CKD-EPI) 6.Clinical status relatively stable 7.Females of childbearing potential must agree to utilize highly effective contraception methods or be non-heterosexually from screening throughout the duration of study treatment and for 30 days following the last dose of study drug.

Exclusion Criteria:

1. A new AIDS-defining condition diagnosed within the 30 days prior to screening
2. Participants experiencing severe organ lesion.
3. Positive serum pregnancy test or planned to be pregnant.
4. Females who are breastfeeding
5. With carcinoma
6. Concomitant medication of immunosuppression or chemoradiotherapy
7. Participation in any other interventional clinical trial
8. Screening stage find: Hb < 9g/dL, WBC < 3000/ul. neutrophilic granulocyte< 1500/ul, PLT< 75000/ul. Scr > 1.5 ULN,Hepatic transaminases (AST and ALT) and ALP > 3 × ULN,total bilirubin ≤ 2 x ULN.
9. Any other clinical condition or prior therapy that, in the opinion of the Investigator, would make the subject unsuitable for the study or unable to comply with dosing requirements

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2021-07-14 (Actual); Primary Completion 2022-12-13 (Actual); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of participants with HIV-1 RNA | base line,Weeks 12,24 and 48
  Proportion of participants with HIV-1 RNA
The Change in CD4 T cell count from baseline | base line,Weeks 12, 24 and 48
  The Change in CD4 T cell count from baseline

CONTACTS AND LOCATIONS:
Overall Officials: Wei Lyu, Principal Investigator — Department of Infectious Diseases, PekingUMCH
Locations (3):
- China (3):
  - The Guangxi Zhuang Autonomous Region Longtan Hospital, Liuchow, Guangxi
  - The Second Hospital of Nanjing, Najing, Jiangsu
  - Tianjin Second People's Hospital, Tianjin